CLINICAL TRIAL: NCT02148601
Title: Fecal Microbiota Transplantation by Colonoscopy for Recurrent C. Difficile Infection: an Open-label Randomized Clinical Trial
Brief Title: Fecal Microbiota Transplantation by Colonoscopy for Recurrent C. Difficile Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Giovanni Cammarota, Prof. Giovanni Cammarota, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A1192013
Record Dates: First submitted 2014-05-23; First posted 2014-05-28 (Estimated); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Clostridium Difficile
Keywords: Fecal microbiota transplantation; Recurrent Clostridium difficile infection; Colonoscopy; Randomized clinical trial
MeSH Terms: conditions — Clostridium Infections | interventions — Fecal Microbiota Transplantation; Vancomycin

ARMS (2):
- Fecal Microbiota Transplantation (Experimental): Fecal microbiota transplantation from healthy donors will be infused by colonoscopy
  Interventions: Other: Fecal Microbiota Transplantation; Drug: Vancomycin (before randomization)
- Standard Antibiotic Therapy (Active Comparator): Standard antibiotic therapy according to European Guidelines (vancomycin and metronidazole) will be administered to the patients
  Interventions: Drug: Standard Antibiotic Therapy; Drug: Vancomycin (before randomization)

INTERVENTIONS:
Other: Fecal Microbiota Transplantation
  Arms: Fecal Microbiota Transplantation
Drug: Standard Antibiotic Therapy
  Arms: Standard Antibiotic Therapy
Drug: Vancomycin (before randomization) — Vancomycin will be administered in all patients for 5 days before randomization. Then, patients will be randomized in FMT Group or Standard Antibiotic therapy Group. Patients in the FMT Group will stop vancomycin 24 hours before the fecal microbiota transplantation. Patients in the Standard Antibiotic Therapy Group will continue vancomycin.

SUMMARY:
In the recent past, a deep change in the epidemiology of C. difficile infection has occurred, with a rise in its frequency, severity, and mortality. Both the refractoriness of the infection to standard therapy and its probability of recurrence have also increased, representing a main clinical issue. Fecal microbiota transplantation (FMT) refers to the introduction of a liquid filtrate of stools from a healthy donor into the gastrointestinal tract of a patient for the treatment of specific diseases. FMT has shown outstanding results in the treatment of recurrent C. difficile infection. It can be performed through various routes: nasogastric or nasojejunal tube, upper endoscopy, retention enema, colonoscopy. In a recent systematic review of studies using FMT for the treatment of recurrent C. difficile infection, Cammarota et al. observed that lower gastrointestinal route (colonoscopy, enema) led to the achievement of higher eradication rates than upper delivery (gastroscopy, naso-gastric or naso-jejunal tube) (81-86% vs 84-93%, respectively). In a randomized clinical trial, Van Nood et al. showed the efficacy of FMT by nasojejunal tube in recurrent C. difficile infection. Up to now, data on FMT by lower route come out only by case series and case reports.

The investigators' aim is to compare the efficacy of colonoscopic FMT and standard antibiotic therapy for the treatment of C. difficile infection in a randomized clinical trial

DETAILED DESCRIPTION:
In the recent past, a deep change in the epidemiology of C. difficile infection has occurred, with a rise in its frequency, severity, and mortality. Both the refractoriness of the infection to standard therapy and its probability of recurrence have also increased, representing a main clinical issue. Fecal microbiota transplantation (FMT) refers to the introduction of a liquid filtrate of stools from a healthy donor into the gastrointestinal tract of a patient for the treatment of specific diseases. FMT has shown outstanding results in the treatment of recurrent C. difficile infection. It can be performed through various routes: nasogastric or nasojejunal tube, upper endoscopy, retention enema, colonoscopy. In a recent systematic review of studies using FMT for the treatment of recurrent C. difficile infection, Cammarota et al. observed that lower gastrointestinal route (colonoscopy, enema) led to the achievement of higher eradication rates than upper delivery (gastroscopy, naso-gastric or naso-jejunal tube) (81-86% vs 84-93%, respectively). In a randomized clinical trial, Van Nood et al. showed the efficacy of FMT by nasojejunal tube in recurrent C. difficile infection. Up to now, data on FMT by lower route come out only by case series and case reports.

The investigators' aim is to compare the efficacy of colonoscopic FMT and standard antibiotic therapy for the treatment of C. difficile infection in an open-label randomized clinical trial The investigators' trial should confirm the clinical results obtained by Van Nood et al. by using a colonoscopy approach.

The investigators' study is an open-label randomized controlled trial, enrolling patients with recurrent C. difficile infection, who are candidates for further antibiotic treatment in accordance with guidelines. Recurrent C. difficile infection is meant as the reappearance of clinical symptoms and positivity of C. difficile toxin test within 8 weeks after the end of the previous therapy. Patients' stool will be screened for detection of parasites and enteric bacterial pathogens to exclude other infective pathogens. Patients with severe clinical features (sepsis, severe dehydration, major co-morbidities), former colectomy, high-risk of endoscopic complications, inflammatory bowel diseases (IBD), irritable bowel syndrome (IBS), viral hepatitis, AIDS or syphilis will be excluded.

Patients will be instructed and invited to signal recurrent symptoms and diarrhea after treatment. Monthly clinical and lab checks will be performed for a period of six months after the treatment.

Treatment procedures:

All patients will start therapy with vancomycin for four days before of stratification, with random allocation (1 to 1) to one of the two treatment schemes: 1) FMT, with the infusion in the cecum - through the biopsy channel - of 60-120 gr (depending on production) of donated feces, obtained from the donor within 6 hours from transplantation, and manually homogenized in 100/200 ml of physiological solution; or 2) standard vancomycin-based therapy according to the international recommendations. Colonoscopy will be performed by an expert endoscopist, with mucosal biopsy (when possible) for histology examination. Patients allocated to FMT arm will undergo preparation for colonoscopy (four liters of a solution with saline laxatives). All patient will be instructed on hygiene rules to be followed at the patient's domicile to avoid re-infections at home. Stool donors should preferably be patient's relatives or intimates, must not have taken antibiotics in the last 6 months, should not present significant intestinal symptoms of other intestinal diseases and must result negative at the serum screening for viral hepatitis, AIDS or syphilis. Their stool will be tested for C. difficile, enteric bacteria, intestinal protozoa and helminthes pathogens.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic recurrent C. difficile infection identified by positivity of C. difficile toxin in stools (ELISA)
* Possibility to undergo standard antimicrobial therapy for recurrent C. difficile infection
* Approval of informed consent
* Possibility to undergo protocol diagnostic and therapeutic procedures
* Stool negativity for parasites
* Stool negativity for Salmonella spp., Shigella spp., Yersinia enterocolitica, Campylobacter, Streptococcus agalactiae, Staphylococcus aureus, enteropathogenic Escherichia coli and other microorganisms except for C. difficile
* Blood negativity for: Hepatitis A virus-Immunoglobulin M, HBsAg, Anti-Hepatitis C Virus, Anti-Human Immunodeficiency Virus1-2, venereal disease reaction level (VDRL).

Exclusion Criteria:

* Subjects <18 years old
* Main comorbidities
* Prior colectomy
* Negativity of C. difficile toxin in stools
* High risk of post-colonoscopy complications
* Other main gastrointestinal diseases (es. Crohn's disease or ulcerative colitis)
* Stool positivity for parasites
* Stool positivity for Salmonella spp., Shigella spp., Yersinia enterocolitica, Campylobacter, Streptococcus agalactiae, Staphylococcus aureus, enteropathogenic Escherichia coli and other microorganisms except for C. difficile
* Blood positivity for: Hepatitis A virus-Immunoglobulin M, HBsAg, Anti-Hepatitis C Virus, Anti-Human Immunodeficiency Virus1-2, venereal disease reaction level (VDRL).
* Pregnancy or breastfeeding.
* Inability to follow protocol procedures

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2013-07; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Disappearance of clinical symptoms linked to C. difficile infection | 10 weeks

SECONDARY OUTCOMES:
Negativization of C. difficile toxin in stools | 10 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of Sacred Heart - "A. Gemelli" University Hospital, Rome, Italy

REFERENCES:
- [Background] Cammarota G, Ianiro G, Bibbo S, Gasbarrini A. Gut microbiota modulation: probiotics, antibiotics or fecal microbiota transplantation? Intern Emerg Med. 2014 Jun;9(4):365-73. doi: 10.1007/s11739-014-1069-4. Epub 2014 Mar 25. PMID 24664520
- [Background] Cammarota G, Ianiro G, Gasbarrini A, Masucci L, Sanguinetti M. Faecal transplantation for Clostridium difficile infection. Three cases treated in Italy. Dig Liver Dis. 2014 May;46(5):475. doi: 10.1016/j.dld.2013.12.011. Epub 2014 Jan 20. No abstract available. PMID 24457126
- [Background] Cammarota G, Ianiro G, Gasbarrini A. Fecal microbiota transplantation for the treatment of Clostridium difficile infection: a systematic review. J Clin Gastroenterol. 2014 Sep;48(8):693-702. doi: 10.1097/MCG.0000000000000046. PMID 24440934